CLINICAL TRIAL: NCT00690625
Title: Topical Application of MyoRx (Omega 3 Fatty Acids Containing) Cream; Randomized Double Blind Clinical Trial
Brief Title: Topical Application of MyoRx (Omega 3 Fatty Acids Containing) Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Ashwini Khante, University Of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-9505-B 01
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Myofacial Pain
Keywords: Myofacial pain; Omega 3 fatty acids
MeSH Terms: conditions — Facial Pain | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): MyoRx cream
  Interventions: Drug: MyoRx Cream (6% Omega 3 Fatty Acid)
- B (Placebo Comparator): Placebo cream, same composition as experimental cream, without Omega 3 fatty acid
  Interventions: Drug: Placebo cream, no Omega 3 fatty acid

INTERVENTIONS:
Drug: MyoRx Cream (6% Omega 3 Fatty Acid) — 1/2 teaspoon 3 times per day for 30 days.
  Arms: A
Drug: Placebo cream, no Omega 3 fatty acid — Placebo cream, no Omega 3 fatty acid
  Arms: B

SUMMARY:
This study is designed to evaluate the effectiveness of topical application of omega-3 fatty acids (6% by volume) containing cream on persons with a TMD disorder, specifically with a diagnosis of Myofacial Pain. Omega-3 fatty acids have minimal side effects when applied topically. If Omega-3 fatty acids used in this study are shown to reduce myofacial pain then this formulation could potentially be used for treatment of TMD patents with myofacial pain in the future. Omega-3 fatty acids are natural ingredients with almost no side effects. Topical application can lead to fewer side effects than systemic medications. In addition, there is no substantial morbidity & mortality associated with topical application of Omega-3 fatty acids. It is hypothesized that subjects receiving topical application of omega-3 fatty acids will demonstrate reduced subjective masseter muscle pain in comparison to subjects receiving placebo cream. This is a pilot study to assess the topical application of Omega-3 fatty acids on muscle pain in the muscles of mastication.

DETAILED DESCRIPTION:
The prevalence of clinically significant temporomandibular disorder (TMD)-related jaw pain has been estimated to be between 3% and 5%. Temporomandibular disorders (TMDs) are a group of conditions characterized by pain or dysfunction in the temporomandibular joint (TMJ), the articular disc and/or the muscles of mastication. TMD is typically classified into three major diagnostic categories, using RDC-TMD classification criteria these would include Myofacial pain (with or without limitation), Disc Displacements (with and without reduction, including with a limited opening,) and Arthralgia, Arthritis and Arthrosis. These pain problems are about twice as common in women as in men in the general population and even four times more common in women in patient populations. A wide range of treatment modalities have been used for the management of myofacial pain. Physical treatments include ultrasound therapy, appliance therapy, intramuscular and nerve root stimulation, anesthetic injection, botulinum toxin injection and dry needling of trigger points, physical therapy, acupuncture and spray and stretch. The major goal of these treatments is to relieve pain and tightness of the involved muscles. Omega-3 fatty acids or fish oil are a family of polyunsaturated fatty acids. Omega-3 fatty acids are powerful anti-inflammatories and lower proinflammatory cytokines. However to obtain any discernible beneficial effects, large doses of Omega-3 fatty acids are required. Thus, topically applied alternatives prove beneficial over systemic routes. Studies show the anti-inflammatory properties of the Omega-3 fatty acids.

This study is designed to evaluate the effectiveness of topical application of omega-3 fatty acids (6% by volume) containing cream on persons with a TMD disorder, specifically with a diagnosis of Myofacial Pain. Omega-3 fatty acids have minimal side effects when applied topically. If Omega-3 fatty acids used in this study are shown to reduce myofacial pain then this formulation could potentially be used for treatment of TMD patents with myofacial pain in the future. Omega-3 fatty acids are natural ingredients with almost no side effects. Topical application can lead to fewer side effects than systemic medications. In addition, there is no substantial morbidity & mortality associated with topical application of Omega-3 fatty acids. It is hypothesized that subjects receiving topical application of omega-3 fatty acids will demonstrate reduced subjective masseter muscle pain in comparison to subjects receiving placebo cream. This is a pilot study to assess the topical application of Omega-3 fatty acids on muscle pain in the muscles of mastication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited who are ages 18 to 70 with a current diagnosis of myofacial pain (using RDC-TMD criteria) including pain on palpation of the masseter muscle. Subjects will be recruited from the Oral Medicine Clinic, School of Dentistry. Because this is a small pilot study, and there will not be sufficient sample size/power, only female subjects will be recruited, as temporomandibular disorder is more prevalent in women than men. Additional inclusion criteria include a "Characteristic Pain Intensity" (CPI) self reported score of three or more. This will be recorded on "Baseline Questionnaire".

Exclusion Criteria:

* Study exclusion criteria:

  1. Males
  2. History of the trauma in last six months
  3. Other chronic pain conditions such as physician diagnosis of fibromyalgia, rheumatoid arthritis, etc
  4. Diagnosis of the disc displacement without reduction with limited opening of TMJ
  5. Age (less than 18 and more than 70)
  6. Evidence of complicating psychological or physical conditions which would prevent the subject from understanding/ participating in the study protocol
  7. Temporomandibular joint surgery on the affected side
  8. Allergy to any of the ingredients in the placebo and the active cream.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the score on the Characteristic Pain Intensity (CPI) scale is 0-10, ordinal. | one month

SECONDARY OUTCOMES:
Secondary outcome measure is satisfaction with the cream, Pain medicine use, | One month

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini V Khante, DDS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Medical center, Department of Oral Medicine, Seattle, Washington, United States